CLINICAL TRIAL: NCT03149393
Title: Clinical Study on Post Evaluation After Listing of Qizhi Weitong Granules
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Digestion-05
Record Dates: First submitted 2017-04-16; First posted 2017-05-11 (Actual); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Functional Dyspepsia; Traditional Chinese Medicine
Keywords: Functional Dyspepsia; Qizhi Weitong Granules; Traditional Chinese Medicine
MeSH Terms: interventions — mosapride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Qizhi Weitong Granules Group (Experimental): Patients in this group will take Qizhi Weitong Granules for 8 weeks.
  Interventions: Drug: Qizhi Weitong Granules
- Mosapride Citrate Tablets Group (Active Comparator): Patients in this group will take mosapride citrate tablets for 8 weeks.
  Interventions: Drug: Mosapride Citrate Tablets

INTERVENTIONS:
Drug: Qizhi Weitong Granules — Patients in this group will take Qizhi Weitong Granules 2.5g,3 times/day,30 minutes before dinner for 8 weeks.
  Other Names: The Treatment Group
  Arms: Qizhi Weitong Granules Group
Drug: Mosapride Citrate Tablets — Patients in this group will take mosapride citrate tablets 5mg,3 times/day,30 minutes before dinner for 8 weeks.
  Other Names: The Control Group
  Arms: Mosapride Citrate Tablets Group

SUMMARY:
This study is a randomized, double blind, double dummy, multicenter, parallel controlled clinical trial, the investigators objective is to evaluate the efficacy and safety of Qizhi Weitong granules in the treatment of functional dyspepsia.

DETAILED DESCRIPTION:
This study is a randomized, double blind, double dummy, multicenter, parallel controlled clinical trial, the investigators objective is to evaluate the efficacy and safety of Qizhi Weitong granules in the treatment of functional dyspepsia. The experiment will be carried out in 8 sub centers at the same time, and the investigators estimated that there will be 384 cases of income, including the experimental group and the control group (n = 192), and the investigators choose mosapride citrate tablets for drug control.

ELIGIBILITY:
Inclusion Criteria:

1. Metting the diagnostic criteria of functional dyspepsia in Rome IV.
2. The subjects were informed, and the subjects voluntarily signed informed consent.
3. The subjects have reading ability.

Exclusion Criteria:

1. Patients suffering from gastric ulcer, gastroscopy see bleeding and mucosal erosion, pathological examination showed atrophy of gastric mucosa, intestinal metaplasia or dysplasia.
2. Patients with Hp infection positive.
3. Patients with gastroesophageal reflux disease.
4. Patients with digestive system organic lesions.
5. The patient had a history of stomach or abdominal surgery.
6. Patients had taken the relevant drugs in the past 2 weeks.
7. Patients suffering from severe illness affecting survival.
8. Pregnant or lactating women.
9. Participating in clinical trials of other drugs.
10. Long term using of sedative hypnotics.
11. Suspected or true alcohol, drug abuse history.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of Main Symptom Score | The score will be assessed at baseline and 2 week, 4 week, 6 week.
  The Main Symptom Score contains evaluation of postprandial fullness discomfort, early satiety, epigastric pain, epigastric burning sensation and so on.

SECONDARY OUTCOMES:
Change of the Hamilton Anxiety Scale and the Hamilton Depression Scale | The score will be assessed at baseline and 2 week, 4 week, 6 week.
  To evaluate the changes of patients' mental and psychological status

CONTACTS AND LOCATIONS:
Overall Officials: Tang X dong, PhD, Study Director — Director of Xiyuan Hospital
Locations (1):
- Xiyuan Hospital, China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No